CLINICAL TRIAL: NCT05156528
Title: A Multicenter, Randomized, Double-blind, Placebo-Controlled Phase III Clinical Trial to Evaluate the Efficacy, Immunogenicity and Safety of S. Flexneriza-S. Sonnei Bivalent Conjugate Vaccine in Volunteers Aged From 6 Months to 5 Years
Brief Title: Efficacy, Immunogenicity and Safety of S. Flexneriza-S. Sonnei Bivalent Conjugate Vaccine in Volunteers Aged From 6 Months to 5 Years
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2021080C
Record Dates: First submitted 2021-12-08; First posted 2021-12-14 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Dysentery; Shigellosis
MeSH Terms: conditions — Dysentery; Dysentery, Bacillary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): S. Flexneriza-S. Sonnei Bivalent Conjugate Vaccine, 0.5ml/dose, 2 doses with an interval of 30 days.
  Interventions: Biological: S. Flexneriza-S. Sonnei Bivalent Conjugate Vaccine
- Placebo group (Placebo Comparator): Aluminium phosphate adjuvant, 0.5ml/dose, 2 doses with an interval of 30 days.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: S. Flexneriza-S. Sonnei Bivalent Conjugate Vaccine — Single intramuscular dose contains 10 µg of S. flexneri 2a polysaccharide and S. sonnei polysaccharide respectively.
  Arms: Experimental group
Biological: Placebo — Single intramuscular dose contains 0.15~0.25 mg of aluminum ion
  Arms: Placebo group

SUMMARY:
The purpose of this study is to evaluate the efficacy, immunogenicity and safety of S. Flexneriza-S. Sonnei Bivalent Conjugate Vaccine in infants and children aged from 6 months to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Infants and children aged from 3 months to 5 years old;
* The legal representative voluntarily agrees to participate in the study and signed the informed consent form;
* The legal representative voluntarily agrees to comply with the requirements of the clinical study protocol, and they can participate in all planned follow-up;
* Subjects who didn't immuned with attenuated live vaccine within 14 days and inactivated vaccine within 7 days before vaccination;
* Axillary temperature ≤37.0℃;
* According to the medical history, physical examination and the judgment of the researcher, it is determined that the subject is in good physical condition.

Exclusion Criteria:

* Previous proven history of bacillary dysentery;
* Subjects who are allergic to tetanus toxoid, and have any history of other vaccination or drug allergy, or a fever above 39.5 ℃ after previous vaccination;
* Within 3 days before vaccination, suffering from acute diseases or in the acute episode of chronic disease or using antipyretic, analgesic and antiallergic drugs (such as acetaminophen, ibuprofen, etc.);
* Had severe bowel disease, and had symptoms such as diarrhea, abdominal pain, pus and blood stool and other symptoms in the past 3 days;
* With pathological jaundice confirmed by existing diagnosis;
* History of thrombocytopenia or other coagulation disorders with definite diagnosis;
* Known or suspected immunological deficiency (such as perianal abscess, which indicates that infants may have immune deficiency), and received long-term (≥14 days) immunosuppressive therapy (radiotherapy, chemotherapy, systemic glucocorticosteroids≥2 mg/kg/day, antimetabolic drugs and cytotoxic drugs) within half a year before vaccination, or confirmed that the parents were HIV infected;
* Received immunoglobulin / blood products treatment within 3 months before vaccination;
* Severe congenital malformations (functional impairment of important organs), severe malnutrition, developmental disorders and serious genetic diseases (such as severe thalassemia);
* Subjects with the following diseases:

  1. Serious liver and kidney diseases, cardiovascular diseases, malignant tumors and other chronic diseases;
  2. Diagnosis with infectious diseases such as tuberculosis, viral hepatitis and so on;
  3. Severe asthma;
  4. Systemic rash, dermatophyte, skin suppuration or blister;
  5. History or family history of convulsion, epilepsy, encephalopathy, mental illness;
* Planning to participate or currently participating in clinical trials of other vaccines or drugs;
* Any situation that the investigator believed may affect the study evaluation.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21000 (Estimated)
Dates: Start 2021-12-11 (Actual); Primary Completion 2024-01-11 (Estimated); Study Completion 2024-01-11 (Estimated)

PRIMARY OUTCOMES:
Efficacy study of S. Flexneriza-S. Sonnei Bivalent Conjugate Vaccine as assessed by protective rate | 30 day after each vaccination
  Evaluate the protective rate for bacillary dysentery

CONTACTS AND LOCATIONS:
Overall Officials: Lin Du, Study Chair — Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd
Locations (9):
- China (9):
  - Hezhou Center for Disease Control and Prevention, Hezhou, Guangxi
  - Luzhai Center for Disease Control and Prevention, Luzhai, Guangxi
  - Sanjiang Center for Disease Control and Prevention, Sanjiang, Guangxi
  - Zhongshan Center for Disease Control and Prevention, Zhongshan, Guangxi
  - Yongnian Center for Disease Control and Prevention, Handan, Hebei
  - Yuanshi Center for Disease Control and Prevention, Huaiyang, Hebei
  - Panzhihua Center for Disease Control and Prevention, Panzhihua, Sichuan
  - Zigong Center for Disease Control and Prevention, Zigong, Sichuan
  - Fushun Center for Disease Control and Prevention, Zigong, Sichuan